CLINICAL TRIAL: NCT02791854
Title: Improving the Quality of Care for Adults With Inflammatory Bowel Disease
Acronym: IBD:QORUS
Status: Enrolling by invitation | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Crohn's and Colitis Foundation (Other); Cedars-Sinai Medical Center (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Corey Siegel, Section Chief, Section of Gastroenterology, Dartmouth-Hitchcock Medical Center
Other Study IDs: OSP#510516 D16124; Award#P01193 (Other: Crohn's and Colitis Foundation)
Record Dates: First submitted 2016-05-13; First posted 2016-06-07 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry participant: This is a registry study, the same information is collected from all participants.

SUMMARY:
Innovative programs exist that suggest that care for people with chronic conditions is optimized when patients and providers have the information they need at the point of care and over time, to engage in shared planning and execution of treatment goals and care plans. This project aims to build an Inflammatory Bowel Disease Learning Health System, a shared information environment, that highlights collaboration among patients, clinicians and care team members, and researchers; for effective use of data for guiding care, value, improvement, and research.

DETAILED DESCRIPTION:
To demonstrate the impact of an Adult Inflammatory Bowel Disease (IBD) Learning Health System approach the study collaborators will design, build, implement, and evaluate in up to 90 IBD care sites the the following four key components of the IBD Learning Health System: 1) a Health Information Technology (HIT) environment that can "feed-forward" Patient Reported Outcomes (PROs) and clinical data to be used at the point of care and integrated into a registry (IBD Plexus); 2) decision-support dashboards for use by patients and clinicians in real time to coproduce care; 3) meaningful reports for patients and clinicians; and 4) multi-stakeholder collaborative networks for improvement and research.

Prior work from Sweden and the US show that successful uptake of the model can offer important benefits. Patients will be able to use web-based tools to monitor their health and manage their care, securely share data with clinicians in a timely manner, visualize outcomes that matter to them, and compare their results to other people. Clinicians will have new information that can improve their ability to track patient outcomes and costs over time; use PRO data to support pre-visit planning, shared decision-making at the point of care, and post-visit monitoring; and receive comparative performance reports to support quality improvement, public reporting, and professional development. Researchers will benefit by having PROs and cost data added to data registries to support clinical, translational, and comparative effectiveness research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of Crohn's disease or ulcerative colitis or IBD unclassified
* Accept the terms and conditions of Informed Consent and Authorization
* Affiliated with a participating IBD Qorus site

Exclusion Criteria:

* Inability to provide informed consent
* Study key personnel cannot enroll as a study participant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In order to participate in IBD Qorus, individuals must meet the following criteria:
  * 18 years of age or older
  * Diagnosis of Crohn's disease or ulcerative colitis or IBD unclassified
  * Accept the terms and conditions of Informed Consent and Authorization
  * Affiliated with a participating IBD Qorus site
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-02-26 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled | annually, up to 5 years
  count of number of patients consented

SECONDARY OUTCOMES:
Proportion of patients in remission | annually, up to 5 years
  assessed using a validated disease activity scale
Proportion of patients on steroids | annually, up to 5 years
  assessed by patient report
Proportion of patients admitted into the Emergency Room | annually, up to 5 years
  assessed by patient report
Proportion of patients hospitalized | annually, up to 5 years
  assessed by patient report
Proportion of patients with anemia | annually, up to 5 years
  assessed by patient report and labs
Proportion of patients with malnutrition | annually, up to 5 years
  assessed by patient report and labs

CONTACTS AND LOCATIONS:
Overall Officials: Corey Siegel, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center; Gil Melmed, MD, MS, Principal Investigator — Cedars-Sinai Medical Center
Locations (29):
- United States (29):
  - Cedars-Sinai Inflammatory Bowel Disease Center, Los Angeles, California
  - Hoag Digestive Health, Newport Beach, California
  - UC San Diego Health Inflammatory Bowel Disease Center, San Diego, California
  - University of Colorado Health, Denver, Colorado
  - Yale School of Medicine IBD Program, New Haven, Connecticut
  - MedStar Georgetown University Hospital Center for Inflammatory Bowel Disease, Washington D.C., District of Columbia
  - Gastro Health LLC, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Digestive Health Center, Boise, Idaho
  - University of Chicago Medicine Inflammatory Bowel Disease Center, Chicago, Illinois
  - Digestive Care Center, Evansville, Indiana
  - GastroIntestinal Specialists, A.M.C., Shreveport, Louisiana
  - Corewell Health, Grand Rapids, Michigan
  - Dartmouth-Hitchcock Inflammatory Bowel Disease Center, Lebanon, New Hampshire
  - Saratoga Schenectady Gastroenterology Associates, Burnt Hills, New York
  - NYU Long Island- Inflammatory Bowel Disease Center, Mineola, New York
  - New York University Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - The Oregon Clinic - Gastroenterology, Portland, Oregon
  - Penn State Hershey Inflammatory Bowel Disease Center, Hershey, Pennsylvania
  - Regional GI, Lancaster, Pennsylvania
  - Gastroenterology Associates, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine IBD Center, Houston, Texas
  - University of Utah Health Care, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided